CLINICAL TRIAL: NCT07105709
Title: A Multi-Centre, Single Arm, Open-Label Extension Study to Evaluate the Long-term Safety and Efficacy of GSK4527226 (AL101) in Participants With Early Alzheimer's Disease
Brief Title: Open-label Extension Study in Participants With Early Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 223646; 2025-521107-42 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2025-08-01; First posted 2025-08-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK4527226 (Experimental): Participants will receive GSK4527226.
  Interventions: Drug: GSK4527226

INTERVENTIONS:
Drug: GSK4527226 — GSK4527226 will be administered.

SUMMARY:
The study medicine GSK4527226 is being studied in participants with Alzheimer's Disease (AD) in study 219867 (the parent study, NCT06079190). This new study is an extension of that parent study called an open-label extension (OLE). An OLE is a clinical trial where all participants receive the same study medicine. Participants must already be in study 219867 to be able to take part in this study. This study will assess the long-term safety and efficacy of GSK4527226 in participants with early AD (including mild cognitive impairment [MCI] and mild dementia due to AD) who have completed the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Treatment Period in the parent study (NCT06079190).
* Participants may have missed doses during the Treatment Period or may be on a temporary dose suspension but must not have been permanently discontinued early from study intervention or withdrawn from the parent study.
* Willing and able to give informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
* Availability of an adult person who has frequent and sufficient contact with the participant, is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits, and signs the study partner ICF.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and if of childbearing potential follows contraception requirements outlined in the protocol.
* A male participant is eligible to participate if he follows contraception requirements outlined in the protocol.

Exclusion Criteria:

* QT interval corrected (QTc) assessment at Day 1 that meets the stopping criteria described in the protocol.
* Participant is taking or will be starting a prohibited medication described in the protocol.
* Evidence of any Amyloid related imaging abnormalities (ARIA) or cerebral macrohemorrhage that meets the permanent discontinuation criteria described in the protocol.
* Other newly identified intracranial hemorrhage aneurysm, vascular malformation, infective lesion, space occupying lesion or brain tumor, or other Magnetic resonance imaging (MRI) findings contraindicating participation in the study.
* Newly identified infection(s) that may affect the Central nervous system (CNS).
* New diagnosis of moderate to severe alcohol and/or substance use disorder.
* Change in participant's ability to tolerate MRI procedures, contraindication to MRI, or any other clinical history or examination finding that would pose a potential hazard in combination with MRI.
* Newly diagnosed cancer.
* Newly identified severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* Newly identified genetic predisposition for clotting disorder or hemorrhagic disease.
* Any other clinically significant change in health status (which, in the opinion of the investigator, would make the participant unsuitable for participation in the OLE study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-12-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) during the OLE | Up to 112 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of Participants with Adverse Event of Special Interest (AESIs) during the OLE | Up to 112 Weeks
  AESIs includes Infusion-related reactions, Amyloid related imaging abnormalities (ARIA) and cerebral macrohemorrhage.
Number of Participants with Serious Adverse Events (SAEs) during the OLE | Up to 112 Weeks
  A SAE is defined as any untoward medical occurrence that, at any dose, results in death and is life threatening requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is a birth defect or congenital anomaly.
Number of Participants with Amyloid related imaging abnormalities (ARIAs) Including Severity during the OLE | Up to 112 Weeks
  Magnetic resonance imaging (MRIs) will be used to monitor for abnormalities in the brain such as brain swelling and/or brain bleeding, which are termed as ARIAs.

SECONDARY OUTCOMES:
Change from OLE Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score Across Weeks 24, 52, 76, and 104 | Baseline, Week 24, 52, 76, and 104
  The CDR-SB score is a quantitative general index that provides more precision in participants with mild dementia. The CDR scale is a clinician-rated dementia staging system tracks the progression of cognitive impairment in 6 categories (memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5- point scale in which 0=None, 0.5=Questionable, 1= Mild, 2=Moderate, and 3=Severe. The CDR-SB score is obtained by adding the ratings in each of the 6 categories and total score ranges from 0 to 18 with higher scores indicative of greater impairment.
Change from OLE Baseline in AD Assessment Scale-Cognitive subscale (ADAS-Cog14) Score Across Weeks 24, 52, 76, and 104 | Baseline, Week 24, 52, 76, and 104
  The AD Assessment Scale-Cognitive subscale (ADAS-Cog14) is a 14-item version of the test that assesses immediate and delayed memory, confrontational naming, ability to follow commands, ideational and constructional praxis, orientation, language, and attention. The ADAS Cog-14 score ranges from 0 to 90 and higher scores indicate greater impairment.
Change from OLE Baseline in Mini - Mental State Exam (MMSE) Across Weeks 24, 52, 76, and 104 | Baseline, Week 24, 52, 76, and 104
  The MMSE is a brief test used to screen for cognitive impairment. It is routinely used for estimating the severity of cognitive impairment and tracking cognitive changes in an individual over time. The MMSE assesses orientation (time and place), registration, attention and calculation, recent memory, language (naming, comprehension, and repetition), and constructional praxis (copying a figure). The MMSE score ranges from 0 to 30, with higher scores indicating better cognitive performance.
Change from OLE Baseline in ADCS-ADL-MCI Score Across Weeks 24, 52, 76, and 104 | Baseline, Week 24, 52, 76, and 104
  The AD Cooperative Study - Activities of Daily Living Scale for use in Mild Cognitive Impairment (ADCS-ADL-MCI). The ADCS-ADL for MCI is a 23-item scale that measures the competence of participants in basic and instrumental activities of daily living. Total scores on the ADCS-ADL-MCI range from 0 to 53 where lower scores indicates greater functional impairment.
Change from OLE Baseline in Integrated Alzheimers Disease Rating Scale (iADRS) Score Across Weeks 24, 52, 76, and 104 | Baseline, Week 24, 52, 76, and 104
  The iADRS is a composite tool that measures both cognition and function. The iADRS combines scores from the ADAS-Cog-14 and the Alzheimer's Disease Cooperative Study-instrumental Activities of Daily Living (ADCS-iADL). The ADAS-Cog-14 is a 14-item version of the test that assesses immediate and delayed memory, confrontational naming, ability to follow commands, ideational and constructional praxis, orientation, language, and attention. The ADCS-iADL is a 23-item scale measuring basic and instrumental abilities in participants with mild to moderate AD. The iADRS score is then computed as the sum of the transformed ADAS-Cog14 and the ADCS-iADL with scores ranging from 0 to 144 and lower scores indicating worse performance.
Change from OLE Baseline in Alzheimers Disease Composite Score (ADCOMS) Across Weeks 24, 52, 76 and 104 | Baseline, Week 24, 52, 76 and 104
  The ADCOMS is a composite score comprising scores from the MMSE, ADAS-Cog14, and CDR-SB. It contains a total of 12 cognitive and functional items, including 4 items from the ADAS-Cog14, 2 items from the MMSE, and 6 items from the CDR-SB. The ADCOMS scores range from 0 to 1.97, with a higher score indicative of greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- United States (9):
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Fairfax, Virginia
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
- Australia (2):
  - GSK Investigational Site, Macquarie Park, New South Wales
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (5):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Oulu, Finland
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
- GSK Investigational Site, Junggu, South Korea
- GSK Investigational Site, Barcelona, Spain
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm
- Taiwan (2):
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taoyuan District
- United Kingdom (3):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf